CLINICAL TRIAL: NCT01630551
Title: Omega-3 Fatty Acid Nutritional Supplementation in the Treatment of Ocular Surface Disease Associated With Intraocular Pressure-Lowering Medications
Brief Title: Omega 3 Supplementation and Ocular Surface Disease in Glaucoma
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No participants enrolled
Sponsor: University of Illinois at Chicago (Other)
Collaborators: American Glaucoma Society (Other)
Responsible Party: Principal Investigator, Ahmad A. Aref, MD, Assistant Professor, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2011-1136
Record Dates: First submitted 2012-05-31; First posted 2012-06-28 (Estimated); Last update posted 2017-02-28 (Actual); Status verified 2017-02

CONDITIONS: Ocular Surface Disease
Keywords: tears; dry eyes; ocular surface disease
MeSH Terms: conditions — Lacerations; Dry Eye Syndromes | interventions — Olive Oil

STUDY DESIGN:
Intervention Model Description: Omega 3 fatty acid
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fishoil nutritional supplement (Active Comparator): 90 day supply of daily oral administration of a fish oil nutritional supplement (TheraTears Nutrition; Advanced Vision Research, Woburn, MA)
  Interventions: Dietary Supplement: Fishoil supplement
- Olive oil capsules (Placebo Comparator): 90 day supply of a daily dose of placebo olive oil capsules
  Interventions: Dietary Supplement: Olive Oil

INTERVENTIONS:
Dietary Supplement: Fishoil supplement — 1 capsule per day
  Arms: Fishoil nutritional supplement
Dietary Supplement: Olive Oil — 1 capsule per day
  Arms: Olive oil capsules

SUMMARY:
Ocular surface disease (OSD) is a significant health problem that affects more than 10 million persons in the United States alone. OSD is highly prevalent among medically treated patients with glaucoma and is associated with the number of intraocular pressure (IOP)-lowering medications used.

The purpose of this study is to determine the potential effectiveness of anoritega-3 fatty acid nutritional supplement in the treatment of ocular surface disease associated"with the use of glaucoma eye drops

DETAILED DESCRIPTION:
Description of procedures/methods:

BASELINE VISIT Once the treating ophthalmologist has made the diagnosis of OSD, subjects will be asked to participate in the research study. Informed consent will be obtained for all subjects willing to participate in the study. Afterwards, the treating ophthalmologist will administer a dry eye questionnaire to each subject. After completion of the questionnaire, subjects will be given 90-day supply of the study drug/placebo. Based on a pre-determined randomization list, each subjects will be randomized to receive either the study medication (TheraTears nutritional supplementation) or a placebo drug (olive oil capsules). All subjects will be instructed to continue using artificial lubrication as needed while taking part in this study.

We hypothesize that therapy with an oral fish oil nutritional supplement containing 450mg EPA, 300 mg DHA, and 1000 mg flaxseed oil (TheraTears Nutrition; Advanced Vision Research, Woburn, MA) will decrease OSD-related symptoms as well as clinical markers associated with OSD (Schirmer test values, positive vital staining with lissamine green, fluorescein tear break-up time, and tear film osmolarity) when compared to administration of placebo.

FOLLOW-UP VISIT Approximately 90 days after the baseline visit, subjects are scheduled to come to the clinic for their routine• eye check. At that visit, subject's O.SD will be re-assessed by the same examination techniques as the baseline visit. After the examination, the questionnaire will be administered for a second time. The study drug will be discontinued at that visit and standard therapy for the subject's OSO, as deemed necessary by the treating ophthalmologist, will be instituted.

Statement of duration of subject participation:

Subject will be in the study for 3 months. There will be two visits, one is the baseline and second is the follow-up visit. All visits will coincide with their regular clinic visit. The total hours of study participation is no more than 2 hours.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Typical symptoms of dry eye (photophobia, burning, foreign body sensation, blurred vision improved with blinking)
* OSDI score > 12
* Schirmer Test with Anesthesia < 8 mm/5 minutes
* Fluorescein tear break-up time < 8 seconds
* No current use of dry eye treatment (except artificial lubrication)

Exclusion Criteria:

* Infectious keratoconjunctivitis or inflammatory disease unrelated to dry eye or topical glaucoma medication use
* Patients with severe tear deficiency (defined as Schirmer tes <5 mm/5 min)
* Concomitant ocular pathology
* History of ocular surgery
* Eyelid or eyelash abnormalities
* Alteration of the nasolacrimal apparatus
* Treatment with drugs affecting tearing
* Treatment with vitamin supplements
* Concomitant ocular therapies
* Topical ophthalmic steroids taken during the 4 weeks before the study
* Pregnant/breast-feeding women
* Women who may be pregnant at the baseline visit or may become pregnant during the 90 days of therapy
* Diabetes
* History of fish and/or shellfish allergy or hypersensitivity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-04; Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Ocular Surface Disease Index Score | 90 Days
  Ocular surface disease validated questionnaire regarding ocular symptoms

SECONDARY OUTCOMES:
Schirmer test score | 90 days
  Scoring of tear production over 5 minutes
Lissamine Green Staining Score | 90 Days
  Ocular staining pattern for significant ocular surface disease
Fluorescein tear break-up time | 90 Days
  Clinical measure of tear film stability

CONTACTS AND LOCATIONS:
Overall Officials: Ahmad A Aref, MD, Principal Investigator — University of Illinois at Chicago College of Medicine
Locations (1):
- Glaucoma Service, Department of Ophthalmology and Visual Science, Chicago, Illinois, United States